CLINICAL TRIAL: NCT00897260
Title: Umbilical Cord Blood Transplantation as Treatment of Adult Patients With Hematologic Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Donna E. Hogge, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H08-02813
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Hematological Malignancy; Bone Marrow Failure Syndrome
Keywords: Unrelated Umbilical Cord Blood Transplant; Multiple cord blood
MeSH Terms: conditions — Hematologic Neoplasms; Bone Marrow Failure Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Umbilical Cord Blood Transplantation as Treatment of Adult Patients with Hematologic Disorders; Radiation: Umbilical Cord Blood Transplantation as Treatment of Adult Patients with Hematologic Disorders; Procedure: Umbilical Cord Blood Transplantation as Treatment of Adult Patients with Hematologic Disorders

INTERVENTIONS:
Drug: Umbilical Cord Blood Transplantation as Treatment of Adult Patients with Hematologic Disorders — To determine the time to and rate of hematologic engraftment following unrelated umbilical cord blood transplantation in adults with one or two cord blood units using total body irradiation and fludarabine as the transplant conditioning regimen and cyclosporine/MMF as graft-versus-host disease prophylaxis.
  DRUG/DOSE DAYS -9 -8, -7 -6 -5 -4 -3 -2 -1 Total Body Irradiation 150 cGy per treatment (1350cGy total) 2x 2x 2x 2x 1x
  * Fludarabine 40mg/m2 10:00am (After TBI) over 60 minutes x x x x Umbilical cord blood infusion (minimum of 24hrs after Flu infusion) x
  * Fludarabine dose adjustment:
    70ml/min: decrease dose by Creatinine Clearance 20% Fludarabine dosing will be based on the 40% adjusted ideal body weight.
  UCB Infusion
Radiation: Umbilical Cord Blood Transplantation as Treatment of Adult Patients with Hematologic Disorders — DRUG/DOSE DAYS -9 -8, -7 -6 -5 -4 -3 -2 -1 Total Body Irradiation 150 cGy per treatment (1350cGy total) 2x 2x 2x 2x 1x
Procedure: Umbilical Cord Blood Transplantation as Treatment of Adult Patients with Hematologic Disorders

SUMMARY:
To determine the time to and rate of hematologic engraftment following unrelated umbilical cord blood transplantation in adults with one or two cord blood units using total body irradiation and fludarabine as the transplant conditioning regimen and cyclosporine/MMF as graft-versus-host disease prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

Patients must have a histologically confirmed diagnosis at The Vancouver General Hospital or the BCCA-Vancouver.

Eligible patients will have one of the following underlying diseases:

* High risk acute lymphoblastic leukemia (ALL) in first complete remission, with high risk being defined by the presence of t(4;11), t(9;22) or t(1;19) or patients presenting with extreme hyperleukocytosis (WBC >100x109/L) or failure to achieve a complete remission after standard induction therapy.
* Acute myeloid leukemia (AML) in first complete remission with high risk cytogenetics or failure to achieve complete remission after standard induction therapy. ALL or AML in second or subsequent remission
* Myelofibrosis with myeloid metaplasia.
* Chronic myeloid leukemia in chronic (failed interferon and/or Gleevec) or accelerated phase.
* Myelodysplastic syndrome with IPSS risk category >Int-1
* Aplastic anemia
* Non-Hodgkin's lymphoma, chronic lymphocytic leukemia or Hodgkin's disease in relapse or second or subsequent remission.
* Multiple Myeloma
* No active central nervous system (CNS) disease.
* No 9/10 or better HLA antigen matched related donor or VUD available.
* The patient's condition precludes waiting to search and find a VUD in the Unrelated Donor Registries
* Acceptance of standard blood product support
* Adequate organ function as defined by current Leukemia/BMT Program of BC standards (Appendix 10.1)
* Karnofsky performance status ≥ 80 (Appendix 10.2)

Exclusion Criteria:

* Active infection
* Pregnancy
* Significant psychiatric disorder
* Progressive disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-05; Primary Completion 2013-01-09 (Actual); Study Completion 2013-01-09 (Actual)

PRIMARY OUTCOMES:
To determine the safety and efficacy of multiple cord blood transplantation in patients with hematological malignancy. | 1 year

SECONDARY OUTCOMES:
To determine the 100-day treatment related mortality (TRM), complete remission rate and the 2-year progression free and overall survival rate for patients under going this treatment. | 100 days
To determine the incidence of grades II-IV and grades III-IV acute GVHD and incidence of limited and extensive chronic GVHD. | 1 year
To measure time to immunologic reconstitution as defined by normal numbers of T and B-cells and normal immunoglobulin synthesis | 1 year
To determine rate of hematologic engraftment following umbilical cord blood transplantation with 1-2 cord blood units using total body irradiation & fludarabine as transplant conditioning regimen & cyclosporine/MMF as graft-vs-host disease prophylaxis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Donna Hogge, Principal Investigator — University of British Columbia - Vancouver Coastal Health Research Institute
Locations (1):
- Vancouver General Hospital, Leukemia/BMT Program of BC, Vancouver, British Columbia, Canada

REFERENCES:
- See also: Related Info — http://www.leukemiabmtprogram.com/